CLINICAL TRIAL: NCT04010396
Title: Clinical and Immunological Patterns of Non-infectious Aortic Graft Inflammation in Bovine vs Non-biological Grafts
Brief Title: Immunological Responses in Bovine vs Mechanical Composite Grafts
Acronym: IRBOcomp
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 24.06.2019 V 1.0
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Immune Defect
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood Samples (1 EDTA + 1 Serum vial)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recipients of Bovine Graft: Recruitment and informed consent procedure for blood sampling to conduct immunological testing. In addition a questionnaire on QOL (SF-12) will be used to evaluate the most actual quality of life of these patients.
  Interventions: Other: Blood sampling
- Recipients of Mechanical Graft: Recruitment and informed consent procedure for blood sampling to conduct immunological testing. In addition a questionnaire on QOL (SF-12) will be used to evaluate the most actual quality of life of these patients.
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Blood sampling: 1 EDTA and 1 Serum vial

SUMMARY:
In the first retrospective part of the study the investigators will conduct a data analysis of patients having received a bovine aortic graft. The investigators will analyze charts and CT / MRI at various time intervals and identify if there are signs of inflammation.

In the second prospective part the investigators will select survivors from the first part with and without inflammation signs. If they consent to participate in the study the investigators will do a blood sampling in order to perform further immunological analysis. Additionally, the investigators will examine their quality of life by QoL SF-12 questionnaire.

DETAILED DESCRIPTION:
Part 1 Retrospective database search on subjects that received a Shelhigh graft (n= 116) and subjects that received a mechanical graft (n=50) in a similar time frame, age, gender, co-morbidities, clinical history.

Analyzing CT or MRI report at following time intervals: 3 - 6 months postoperatively, 1, 2 and 3 years postoperatively (regular check-up appointments in clinics).

Additionally, extraction of following data-set (based on availability): temperature, lab values (C-reactive protein, white blood count, Eosinophil count), pathology report and CT- / MRI- imaging in cases of re-operation.

Firstly, identify if there is a graft inflammation (positive / negative group within the bovine group).

Secondly, compare to mechanical group.

Part 2 Choose 10 + 10 patients of the bovine group (with / without immune response) and 10 of the mechanical group in order to conduct further immunological testing and comparison. The immunological testing will include measurement of immunoglobulin E and immunoglobulin G antibodies against bovine protein, as well as in vitro T cell reactivity in Interleukin 4 and interferon-gamma Elispot. These parameters will characterize whether the patient mounted an adaptive immune response against the bovine protein. In addition, the investigators will measure total immunoglobulin G4 and Interleukin-6 levels in the serum of all patients, as additional inflammation markers.

Contact patients to come into clinics for a visit, explain study. Blood sampling (1 serum and 1 EDTA) after patients consent.

Material will be sampled and sent in anonymized form via express courier to the Translational Immunology Lab at the University Hospital Basel. Samples will be processed within 24h to isolate peripheral blood mononuclear cells (PBMC) and serum. PBMC and Serum will be cryopreserved at -180°C and -80°C respectively. Samples will be analyzed in batches each including 3-5 subjects per group.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of the bovine graft or mechanical graft. For the prospective part 2: able to give informed consent by signature, age, matching characteristics and time frame.

Exclusion Criteria:

* Individuals of the patient cohort from the last 20 years who indicated that their data cannot be utilized for future research will be excluded from the study.
* Inability or any contraindications to undergo the planned investigated intervention, clinically significant concomitant diseases precluding ambulatory control in the day clinic in Bern.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Part 1: n=116 bovine (total amount of recipients of the Shelhigh graft at the investigators' institution).
  50 (mechanical control)
  Part 2: n= 10 (bovine with immune response) +10 (bovine without immune response) +10 (mechanical control)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Inflammatory Response | postoperatively, up to 30 years
  Percentage of patients having received the bovine conduit graft showing a graft inflammation.

SECONDARY OUTCOMES:
Inflammatory Response in Control Group | postoperatively, up to 30 years
  Comparison of the bovine group to patients having received a mechanical composite graft.

CONTACTS AND LOCATIONS:
Overall Officials: ThierryThierry Prof. Dr. med. Carrel, Study Chair — Department Chair
Locations (1):
- University Hospital Bern, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrel TP, Schoenhoff FS, Schmidli J, Stalder M, Eckstein FS, Englberger L. Deleterious outcome of No-React-treated stentless valved conduits after aortic root replacement: why were warnings ignored? J Thorac Cardiovasc Surg. 2008 Jul;136(1):52-7. doi: 10.1016/j.jtcvs.2007.09.047. Epub 2008 May 27. PMID 18603053
- [Background] Carrel T, Reineke D, Englberger L. Another report on unfavourable long-term outcome following implantation of the Shelhigh No-React valved tube graft. Eur J Cardiothorac Surg. 2016 Dec;50(6):1179-1180. doi: 10.1093/ejcts/ezw205. Epub 2016 Jun 14. No abstract available. PMID 27307482
- [Background] Reineke DC, Kaya A, Heinisch PP, Oezdemir B, Winkler B, Huber C, Heijmen RH, Morshuis W, Carrel TP, Englberger L. Long-term follow-up after implantation of the Shelhigh(R) No-React(R) complete biological aortic valved conduit. Eur J Cardiothorac Surg. 2016 Jul;50(1):98-104. doi: 10.1093/ejcts/ezv452. Epub 2015 Dec 30. PMID 26719402
- [Background] Gisler F, Huber C, Wenaweser P, Carrel T. Severe calcification of a Shelhigh stentless valved conduit. Eur J Cardiothorac Surg. 2014 Aug;46(2):334. doi: 10.1093/ejcts/ezt569. Epub 2013 Dec 11. No abstract available. PMID 24335263
- [Background] Schoenhoff FS, Loup O, Gahl B, Banz Y, Pavlovic M, Pfammatter JP, Carrel TP, Kadner A. The Contegra bovine jugular vein graft versus the Shelhigh pulmonic porcine graft for reconstruction of the right ventricular outflow tract: a comparative study. J Thorac Cardiovasc Surg. 2011 Mar;141(3):654-61. doi: 10.1016/j.jtcvs.2010.06.068. Epub 2011 Jan 20. PMID 21255796
- [Background] Carrel TP. Another disastrous outcome following aortic root replacement with the Shelhigh No-react aortic valved tube. Thorac Cardiovasc Surg. 2008 Aug;56(5):314-5. doi: 10.1055/s-2008-1038472. No abstract available. PMID 18615385
- [Background] Englberger L, Noti J, Immer FF, Stalder M, Eckstein FS, Carrel TP. The Shelhigh No-React bovine internal mammary artery: a questionable alternative conduit in coronary bypass surgery? Eur J Cardiothorac Surg. 2008 Feb;33(2):222-4. doi: 10.1016/j.ejcts.2007.11.006. Epub 2007 Dec 20. PMID 18083039
- [Background] Sahin A, Muggler O, Sromicki J, Caliskan E, Reser D, Emmert MY, Alkadhi H, Maisano F, Falk V, Holubec T. Long-term follow-up after aortic root replacement with the Shelhigh(R) biological valved conduit: a word of caution! Eur J Cardiothorac Surg. 2016 Dec;50(6):1172-1178. doi: 10.1093/ejcts/ezw167. Epub 2016 May 26. PMID 27229673
- [Background] Kaya A, Heijmen RH, Kelder JC, Schepens MA, Morshuis WJ. Stentless biological valved conduit for aortic root replacement: initial experience with the Shelhigh BioConduit model NR-2000C. J Thorac Cardiovasc Surg. 2011 May;141(5):1157-62. doi: 10.1016/j.jtcvs.2010.07.009. Epub 2010 Sep 15. PMID 20832085